CLINICAL TRIAL: NCT03599388
Title: Extending Sleep to Reverse Metabolic Syndrome in Middle-aged Adults: Acceptability and Feasibility of a Sleep Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-00396
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Sleep; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SASI (Experimental): * Sleep Diaries (daily)
  * Fitbit 24/7
  * Phone/videoconference (weekly with study team)
  * Epworth Sleepiness Scale (weekly)
  * PROMIS fatigue scale-morning (weekly)
  * PROMIS fatigue scale-evening (weekly)
  Interventions: Behavioral: Self- management for adequate sleep intervention (SASI)

INTERVENTIONS:
Behavioral: Self- management for adequate sleep intervention (SASI) — Bedtimes and wake times will be prescribed each week for each participant and allow for gradual increases in sleep opportunity. Bedtimes will be set 15 minutes earlier each week provided sleep efficiency remains >90%. Earlier betimes will extend sleep duration by increasing the opportunity for sleep. Wake times will not be changed because wake times are often determined by external demands, such as work schedules

SUMMARY:
This pilot study will test acceptability and feasibility of a sleep extension intervention in community dwelling, short sleeping, racially/ethnically diverse middle aged adults with Metabolic Syndrome (METs). Baseline sleep habits will be assessed and used to guide individualized strategies to extend sleep. A 1-group pre-test, post-test study design will test the efficacy of this 18 week study (2 weeks of baseline data collection, 1 week of study intervention planning, 12 weeks of sleep intervention planning, 12 weeks of sleep intervention delivery, final follow up 3 weeks after last day of the 12 week intervention) on sleep duration, MetS factors (waist circumference, blood pressure, fasting glucose, trigycerides, HDL-c), MetS risk behaviors (poor affective well-being, fatigue) and self regulation. Socio-ecological barriers and facilitators to the intervention will be identified using a quantitative and qualitative approach.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 40 years of age and less than or equal to 60 years of age.
* Objectively confirmed MetS defined by three or more of the following:

  1. waist circumference greater than 120cm (men) or 88cm (women),
  2. blood pressure greater than or equal to 135 mmHg systolic or greater than or equal to 85 mmHg diastolic or antihypertensive medication use,
  3. fasting glucose greater than or equal to 110 mg/dL or insulin or oral hypoglycemic medication use,
  4. serum triglycerides greater than or equal to 150mg/dL or hypertriglyceridia medication use,
  5. HDL-c less than 40mg/dL (women) or less than 50 mg/dL (men) or medication use for low HDL-c1. MetS was selected because individuals with MetS are at high risk for multiple chronic conditions35.
* No obstructive sleep apnea.
* Accelerometry confirmed short sleep (average work day sleep less than or equal to 6 hours/night).
* English speaking.

Exclusion Criteria:

* Pregnancy/lactation
* Current chemotherapy treatments
* Alcohol abuse/dependence
* Night shift or shift work (previous 2 months)
* trans-meridian travel (previous 4 weeks),
* planned shift work or trans-meridian travel during intervention period
* Insomnia
* Moderate-severe or severe depression
* Sleep-promoting medications
* Habitual napping, defined as 2 naps per day or > 90 minutes of napping on 3 or more days of the week.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Measure of acceptability Pre-Intervention evaluated by the percentage of participants rating SASI as acceptable, neutral, unacceptable | 0 Months
  Acceptable (overall acceptability survey scores greater than 21), neutral (overall acceptability survey scores equal to 21), and unacceptable (overall acceptability survey scores less than 21) at each of two time points
Measure of acceptability Post Intervention evaluated by the percentage of participants rating SASI as acceptable, neutral, unacceptable | 4 Months
  Acceptable (overall acceptability survey scores greater than 21), neutral (overall acceptability survey scores equal to 21), and unacceptable (overall acceptability survey scores less than 21) at each of two time points (pre- intervention and post intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Malone, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose